CLINICAL TRIAL: NCT01804062
Title: Evaluation of Respiration Rate Parameters in Healthy Volunteers Using a Nellcor Bedside Respiratory Patient Monitoring System With Respiration Rate Version 2.0
Brief Title: Respiration Rate V2.0 in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0394
Record Dates: First submitted 2013-02-20; First posted 2013-03-05 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Focus of the Study is Measuring Respiratory Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: no treatment, prospective observational

SUMMARY:
The purpose of this study is to meet the respiration rate accuracy specifications for the study pulse oximeter monitoring system (study device)in a healthy volunteer population when compared to established technologies for measuring parameters related to respiration, such as Capnograph Respiration Rate (RR) (CO2).

DETAILED DESCRIPTION:
Volunteer subjects with no significant medical problems (see specific inclusion/exclusion criteria) over the age of 18, male and female, who provide written informed consent prior to the procedure, are not pregnant, and without any contact skin allergies to adhesives found in standard pulse oximetry sensors.

The study consists of measuring parameters related to respiration in healthy volunteers by means of the Bedside Respiratory Patient Monitoring System with RR V2.0 (Nightingale). The prototype Nightingale device and multiparameter reference devices will be attached to the subject via sensors, nasal cannulas and ECG leads and the information from all devices will be captured continuously for up to 40 minutes to allow for at least 30 minutes of artifact free data 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects.
* 18 years or older.
* Subject is willing and able to provide written consent.

Exclusion Criteria:

* Subject is younger than 18.
* Subject is pregnant or lactating
* Subject has severe contact allergies that may cause a reaction to standard adhesive materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors.
* Subject has an abnormality that may prevent proper application of the device.
* Subject is in atrial fibrillation.
* Subject has a documented history of frequent premature ventricular contractions (PVCs), defined as greater than 3 in 30 seconds or greater than 6 in 60 seconds
* Subject has an implanted pacemaker.
* Subject is unwilling or unable to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer subjects with no significant medical problems
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Kelley, MD, Principal Investigator — Medtronic - MITG
Locations (1):
- Boulder In-House Clinical Laboratory, Boulder, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | no Treatment
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | no Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Error (ME) +/- 1 Breath Per Minute, RR Sensor
Description: The software shall calculate respiration rate values via Adult Respiratory Sensor with a mean error of +/- 1 breath per minute relative to a capnography based reference.
Time Frame: up to 40 minutes of continous monitoring
Measure: Mean (Standard Deviation); unit: BrPM
Arm/Group | no Treatment
Number analyzed (Participants) | 30
BrPM | -0.05 (1.04)

2. Secondary Outcome: ME +/- 1 Breath Per Minute, Max-N Sensor
Description: The software shall calculate respiration rate values via Max-N with a mean error of +/- 1 breath per minute relative to a capnography based reference.
Time Frame: up to 40 minutes of continuous monitoring
Measure: Mean (Standard Deviation); unit: BrPM
Arm/Group | no Treatment
Number analyzed (Participants) | 30
BrPM | -0.03 (1.05)

ADVERSE EVENTS:
Arm/Group | no Treatment
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No